CLINICAL TRIAL: NCT04886765
Title: A Phase I/II, Multi-center, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of ALMB-0168 in Patients With Osteosarcoma
Brief Title: A Study to Evaluate the Safety and Efficacy of ALMB-0168 in Patients With Osteosarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlaMab Therapeutics (Shanghai) Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALMB-0168-CN-101
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALMB-0168 (Experimental): Dose Escalation Cohort ：The accelerated titration and traditional "3+3" design will be used in the dose-escalation phase. Seven dose cohorts will be evaluated. ALMB-0168 will be administered intravenously once every 3 weeks until either the disease progresses or intolerable toxicity occurs.
  Dose Expansion Cohort: Based on the results of Part I, 1-3 dose expansion cohorts will be started to further evaluate the safety and efficacy of ALMB-0168.
  Interventions: Drug: ALMB-0168

INTERVENTIONS:
Drug: ALMB-0168 — ALMB-0168 will be administered intravenously until either the disease progresses or intolerable toxicity occurs.

SUMMARY:
This is a phase I / II, multi-center, single-arm, open-label study to evaluate the safety and efficacy of ALMB-0168 in patients with osteosarcoma whose prior standard treatment have failed.

DETAILED DESCRIPTION:
This is a phase I / II, multi-centre, single-arm, open-label study with two parts, a dose-escalation phase (Part I) and a dose-expansion phase (part II). In part I, patients with osteosarcoma whose prior standard treatment have failed will be assigned to receive sequentially higher doses of ALMB-0168 intravenously. The dose-escalation initially will follow an accelerated titration design for the first two dosing groups, then follow a classic 3+3 design. The maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of ALMB-0168 will be determined in part I. In Part II, 1-3 expansion cohorts will begin to further assess the safety profile and explore efficacy, and each cohort will enroll up to 60 patients with high-grade osteosarcoma in each cohort. All patients will receive multiple administration of ALMB-0168 until either the disease progresses or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed osteosarcoma;
2. Patients will be enrolled according to different stages:

   1. Part I: Patients with osteosarcoma whose prior standard treatment have failed.;
   2. Part II: Patients with high-grade osteosarcoma whose prior standard treatment have failed.; Standard treatment failure is defined as the progression on or within 6 months after the first-line chemotherapy (including high-dose methotrexate, doxorubicin, cisplatin, ifosfamide, etc.); For patients with disease progression more than 6 months after the chemotherapy, the risk-benefit assessment should be conducted by the investigators;
3. 16 years of age or older, male or female;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2;
5. Either measurable or non-measurable disease per RECIST v1.1. Non-measurable disease should be assessable by conventional imaging techniques including isotope bone scans, CT or MRI scans. Patients in part II stage must have at least one measurable lesion confirmed by CT or MRI at baseline.
6. Adequate major system function defined as:

   1. Bone marrow reserve: Absolute neutrophil count (ANC) ≥1.5 x109/L; Platelet count ≥ 75 x 109/L; Hemoglobin ≥ 90 g/L (not receiving blood transfusion within 14 days before the first administration);
   2. Hepatic function: Total bilirubin ≤1.5 x upper limit of normal (ULN), Transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and/or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT)) ≤ 3 x ULN (<5 x ULN for liver metastases);
   3. Renal function: Normal serum creatinine ≤1.5 mg/dL (133 μmol/L) OR calculated creatinine clearance ≥50 mL/min. (Cockcroft - Gault formula);
   4. Coagulation: Adequate coagulation parameters defined as International Normalization Ratio (INR) ≤2.
7. Female patients of childbearing potential must have negative results of serum pregnancy test within 7 days before the first dose. Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including 1 barrier method, during their participation in the study and for 3 months following the last dose. Male patients must also refrain from donating sperm during their participation in the study;
8. Life expectancy ≥3 months;
9. Ability to understand the entire process of this study, voluntarily participate and sign a written informed consent form.

Exclusion Criteria:

1. Any recent anti-tumour therapy ≤ 28 days before the first dose or residual more than Grade 1 chemotherapy-related side effects per NCI CTCAE v5.0, with the exception of alopecia.
2. Have participated in the other clinical trial and received the investigational drug treatment within 4 weeks before the first dose of study drug;
3. Wide-field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy;
4. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement;
5. Brain metastases, leptomeningeal metastases or, spinal cord compression or central nervous system (CNS) injuries/abnormalities;
6. Pregnant women. Breastfeeding women should stop breastfeeding before signing the informed consent;
7. Any of the following cardiac diseases currently or within the last 6 months:

   1. Left ventricular ejection fraction (LVEF) <45% as determined by echocardiogram (ECHO);
   2. The corrected QT interval (Fridericia formula) interval (QTcF) > 470 msec for females and > 450 msec for men in electrocardiogram (ECG) at screening;
   3. Unstable angina pectoris;
   4. Heart failure (New York Heart Association (NYHA) >2 grade);
   5. Acute myocardial infarction;
   6. Uncontrolled arrhythmia;
   7. Acute coronary syndromes;
   8. Stent placement;
8. Uncontrolled hypertension (systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg (Patients with blood pressure values higher than these levels must use drugs to control blood pressure below this level before the first dose of study drug));
9. Have a serious active infection (systemic intravenous antibiotics within 14 days but oral antibiotics allowed) that is not well controlled, or have another serious underlying medical condition that would prevent the patients from receiving the protocol treatment;
10. Known diagnosis of human immunodeficiency virus, active hepatitis B or C;
11. Have received Chinese herbal medicine or Chinese patent drug with anti-tumor activity within 14 days before the first administration;
12. Has other active tumors or a history of infiltrative tumor treatment within 3 years. Patients with a history of definitively locally treated stage I tumors who are considered unlikely to recur can be accepted. Patients with a history of prior treatment for carcinoma in situ (e.g., non-invasive) and history of non-melanoma skin cancer are acceptable.
13. According to the researchers' judgment, patients with other factors that may lead to the termination of the study, such as other serious diseases (including severe mental disorders) requiring combined treatment, serious laboratory abnormalities, family or social factors, which may affect the safety or the collection of data and samples. Psychological, family, social or geographical conditions and other factors are not consistent with the experimental scheme.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From enrollment to 28 days after the last dose in each part study.
  Defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0). Incidence of adverse events will be assessed in both PART I and PART II.
Dose-Limited Toxicities (DLT) | Up to 21 days in Cycle 1
  DLTs were assessed according to NCI-CTCAE v.5.0 during the first cycle
6-Month Progression-free Survival Rate (6m-PFSR) | From enrollment to 6 month after the first dose of the last patient in PART II
  6m-PFSR is defined as the percentage of patients who will be alive and without PD at 6 months from the randomization date. 6m-PFSR will be assessed only in PART II.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  Measure the maximum (peak) plasma concentration
Time to maximum concentration (Tmax) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  Measure the time to reach maximum (peak) plasma concentration
Minimum concentration(Cmin) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  Measure the minimum (trough) plasma concentration
The area under the curve (AUC) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  Measure the area under the curve
Half-life (t1/2) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  calculate the half-life of ALMB-0168
Clearance (CL) of ALMB-0168 | From enrollment to 4 weeks after the last dose of the last patient
  Measure apparent total clearance(s) from plasma after administration
Objective Response Rate (ORR) | 2 year
  ORR will be assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1.
Disease control rate (DCR) | 2 year
  DCR will be determined by Response evaluation criteria in solid tumours v1.1
Duration of response (DOR) | 2 year
  DOR was defined as the time from first documented evidence of complete response (CR) or partial response (PR) until progressive disease (PD) or death.
Progression-free survival (PFS) | up to 3 years
  PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first.
Time to Response (TTR) | 2 year
  TTR was defined as the time to a confirmed CR (disappearance of all target lesions) or PR (At least a 30 percent decrease in the sum of diameters of target lesions) per RECIST 1.1.
Overall survival (OS) | up to 3 years
  OS was defined as the time from randomization to death due to any cause.
Rate of Skeletal Related Events (SRE) | through study completion, an average of 3 year
  Including pathological fractures, spinal cord compression, hypercalcemia caused by malignant tumors, radiotherapy or surgery for bone lesions for symptom relief
Change from baseline in alkaline phosphatase (ALP) and lactate dehydrogenase (LDH) | through study completion, an average of 3 year
  pre- and post-treatment ALP and LDH changes in blood samples
Change from baseline in Bone Mineral Density (BMD) | through study completion, an average of 3 year
  Dual-energy X-ray absorptiometry (DXA) to determine the bone mineral density of the subjects' lumbar spine, hip bone and femoral neck.
Dose of morphine compared with baseline | through study completion, an average of 3 year
  pre- and post-treatment dose changes of morphine
Frequency of morphine compared with baseline | through study completion, an average of 3 year
  pre- and post-treatment frequency changes of morphine
Change from baseline of numeric pain scale (NRS) scores | through study completion, an average of 3 year
  pre- and post-treatment changes of NRS scores (min~max: 0~10; higher scores means a worse outcome)
Change from baseline of quality of life scale (EQ-5D) scores | through study completion, an average of 3 year
  pre- and post-treatment changes of EQ-5D scores (min~max: 0~100; higher scores means a better outcome)
The incidence of anti-drug antibody (ADA) | From enrollment to 4 weeks after the last dose of the last patient
  The percentage of patients with ADA

CONTACTS AND LOCATIONS:
Overall Officials: Jingnan Shen, Doctor, Principal Investigator — the first affiliated Hospital, Sun Yat-sen Unibersity

IPD SHARING:
Plan to Share IPD: No